CLINICAL TRIAL: NCT01058434
Title: A Phase II, Multi-center, Non-randomized, Open-label Study of TKI258 in Patients With Relapsed or Refractory Multiple Myeloma, Who Are With or Without t(4;14) Translocation
Brief Title: Safety and Efficacy of TKI258 in Relapsed or Refractory Multiple Myeloma Patients, Who Are With or Without t(4;14) Chromosomal Translocation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CTKI258A2204; 2009-012417-22 (EudraCT Number)
Record Dates: First submitted 2010-01-26; First posted 2010-01-28 (Estimated); Last update posted 2020-12-19 (Actual); Status verified 2020-08

CONDITIONS: Relapsed or Refractory Multiple Myeloma
Keywords: Multiple myeloma; relapsed; refractory; t(4;14); FGFR3
MeSH Terms: conditions — Recurrence; Multiple Myeloma | interventions — 4-amino-5-fluoro-3-(5-(4-methylpiperazin-1-yl)-1H-benzimidazol-2-yl)quinolin-2(1H)-one

ARMS (1):
- TKI258 (Experimental)
  Interventions: Drug: TKI258

INTERVENTIONS:
Drug: TKI258

SUMMARY:
This study will evaluate safety and efficacy of TKI258 in patients with relapsed or refractory multiple myeloma

ELIGIBILITY:
Inclusion Criteria:

1. Cytopathologically or histologically confirmed diagnosis of multiple myeloma previously requiring systemic treatment.
2. Evidence of relapsed or refractory disease as documented from the prior treatment history. (Refractory myeloma is defined as disease that is non-responsive while on salvage therapy, or progresses within 60 days of last therapy. Relapsed myeloma is defined as previously treated myeloma which after a period of being off-therapy requires the initiation of salvage therapy. Detailed definitions provided in the PTS-1)
3. Have received at least 2 prior treatment regimens for multiple myeloma including chemotherapy, autologous transplantation, immunotherapy, or other investigational agents. Pre-planned induction, followed by transplant and maintenance should be considered as one regimen.
4. Presence of measurable disease as defined by at least one of the following;

   * Serum M-protein ≥ 1g/dL (measurable disease)
   * Urine M-protein ≥ 200mg/24 hours by protein electrophoresis (measurable disease)

Exclusion Criteria:

1. Patients with non-secretory, or oligosecretory, multiple myeloma.
2. Patients with symptomatic amyloidosis, or with plasma cell leukemia.
3. Patients who have received allogeneic stem cell transplantation and who show evidence of active graft-versus-host disease that requires immunosuppressive therapy.

Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2010-05; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Overall response rate | 4 weeks

SECONDARY OUTCOMES:
frequency and severity of adverse events as per CTCAE | throughout the study
Progression free survival (PFS) | every 4 weeks
Plasma exposure of TKI258 | during the first 3 cycles

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (29):
- United States (15):
  - University of South Alabama / Mitchell Cancer Institute Dept. of Mitchell Cancer Inst., Mobile, Alabama
  - Central Hematology Oncology Medical Group, Alhambra, California
  - Central Coast Medical Oncology Corporation, Santa Maria, California
  - St. Jude Heritage Medical Group Virginia Crosson Cancer Center, Yorba Linda, California
  - Kootenai Medical Center Kootenai Medical Center, Coeur d'Alene, Idaho
  - Hematology and Oncology Specialists Dept of Hem&Onc Specialist - 2, Metairie, Louisiana
  - Mayo Clinic - Rochester Rochester, Rochester, Minnesota
  - Memorial Sloan Kettering Cancer Center MSKCC, New York, New York
  - Duke University Medical Center Dept. of DUMC (4), Durham, North Carolina
  - Lancaster Cancer Center, Lancaster, Pennsylvania
  - Cancer Centers of the Carolinas Dept. of CC of the Carolinas, Greenville, South Carolina
  - University of Tennessee Cancer Institute SC-2, Memphis, Tennessee
  - University of Texas Southwestern Medical Center UTSW Medical Center, Dallas, Texas
  - University of Wisconsin SC, Madison, Wisconsin
  - Medical College of Wisconsin Med College of Wisconsin, Milwaukee, Wisconsin
- Australia (3):
  - Novartis Investigative Site, Adelaide, South Australia
  - Novartis Investigative Site, Melbourne, Victoria
  - Novartis Investigative Site, Prahran, Victoria
- Canada (2):
  - Novartis Investigative Site, Toronto, Ontario
  - Novartis Investigative Site, Montreal, Quebec
- Novartis Investigative Site, Nantes, France
- Germany (3):
  - Novartis Investigative Site, Bochum
  - Novartis Investigative Site, Cologne
  - Novartis Investigative Site, Heidelberg
- Netherlands (2):
  - Novartis Investigative Site, Amsterdam
  - Novartis Investigative Site, Rotterdam
- Turkey (Türkiye) (3):
  - Novartis Investigative Site, Altunizade
  - Novartis Investigative Site, Ankara
  - Novartis Investigative Site, Izmir

REFERENCES:
- [Result] Scheid C, Reece D, Beksac M, Spencer A, Callander N, Sonneveld P, Kalimi G, Cai C, Shi M, Scott JW, Stewart AK. Phase 2 study of dovitinib in patients with relapsed or refractory multiple myeloma with or without t(4;14) translocation. Eur J Haematol. 2015 Oct;95(4):316-24. doi: 10.1111/ejh.12491. Epub 2015 Jan 22. PMID 25402977
- See also: CTKI258A2204 Results at Novartis Clinical Trials Results Website — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=9317